CLINICAL TRIAL: NCT00539422
Title: Role of Cytochrome P450 2D6 (CYP2D6) *4 Polymorphism, Oxidative Stress and Ferretin in Benign and Malignant Breast Diseases
Brief Title: Role of Cytochrome P450 2D6 (CYP2D6) *4 Polymorphism,in Malignant Breast Diseases
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Other Study IDs: Role of cytochrome P450 2D6
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; cytochrome 450; CYP2D6*4; Ferritin; oxidative stress; cancer; cancer breast
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Polymerase Chain Reaction; Biomarkers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- I: group I of 15 women with benign breast lesion
  Interventions: Genetic: pcr and serum markers for breast cancer
- II: group II of 16 women with breast cancer
  Interventions: Genetic: pcr and serum markers for breast cancer
- III: 13 women were taken as a control group
  Interventions: Genetic: pcr and serum markers for breast cancer

INTERVENTIONS:
Genetic: pcr and serum markers for breast cancer — DNA extraction and genotyping of cytochrome P450-2D6*4 gene using conventional PCR followed by restriction enzyme (Mva1) digestion. Separated plasma was used for measurement of plasma malondialdehyde(MDA)concentration, total plasma antioxidant capacity and plasma ferretin level.

SUMMARY:
The aim of our study is to investigate the potential role of the CYP2D6*4 polymorphism in breast cancer and furthermore to assess the role of oxidative stress, antioxidant capacity and ferretin in pathogenesis of breast cancer in different CYP2D6*4 genotypes

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among women and the second highest cause of cancer death. Nevertheless most of the breast cancer is sporadic with no family history of the disease, Enhanced CYP2D6 activity has been related to malignancies of the bladder, liver, pharynx, and stomach and, especially, to cigarette-smoking-induced lung cancer. Data support that increased formation of reactive oxygen species (ROS) may play an important role in carcinogenesis Numerous in vitro experiments show that ROS damages DNA, inducing premutagenic modifications of nucleotides and promoting oxidation of proteins and lipid per oxidation The aim of our study is to investigate the potential role of the CYP2D6*4 polymorphism in breast cancer and furthermore to assess the role of oxidative stress, antioxidant capacity and ferretin in pathogenesis of breast cancer in different CYP2D6*4 genotypes.patients and methods : This study included 31 women admitted to the general surgery department, Mansoura University Hospital. group I consists of 15 women with benign breast lesion, group II composed of 16 women with cancer breast and 13 healthy women with matched age and clinically free were taken as a control group. DNA extraction and genotyping of cytochrome P450-2D6*4 gene using conventional PCR followed by restriction enzyme (Mva1) digestion. Separated plasma was used for measurement of plasma malondialdehyde(MDA)concentration, total plasma antioxidant capacity and plasma ferretin level.Results homozygous genotype of 2D6*4 represent 56.25 %( 9/16) of breast cancer group with lower wild type (31.25%-5/16), while it represent 33.3 %( 5/15) of begnine breast lesion group and 15.3(2/13) of the control group. Where the wild type represent the majority of cases (61.15%-8/13) in the control group and 46.6%-7/15) in the begnine breast lesion group.

statistically significant increase in plasma ferretin and MDA mean levels in breast cancer group than begnine breast lesion and the control groups .Also, there is an increase in plasma total antioxidant activity in breast cancer group than the control group with nonstatistical difference between the breast cancer and the benign breast lesion groups .

Conclusion CYP2D6*4 genotype polymorphism interacting with plasma malondialdehyde (MDA) oxidative stress and plasma ferretin level may have a role in the pathogenesis of breast cancer

ELIGIBILITY:
Inclusion Criteria:

* This study included 31 women admitted to the general surgery department, Mansoura University Hospital. group I consists of 15 women with benign breast lesion, group II composed of 16 women with cancer breast and 13 healthy women with matched age and clinically free were taken as a control group.

Ages: 33 Years to 63 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-01; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: wagih m ghnnam, Principal Investigator — mansoura faculty of medicine general surgery department; Aymen z El Samanoudy, Study Director — mansoura faculty of medicine biochemistry department
Locations (1):
- Mansoura Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt